CLINICAL TRIAL: NCT02054078
Title: Efficacy and Safety of Intrapleural Bevacizumab Versus Pulvis Talci in Malignant Pleural Effusion, A Randomized, Multicenter Study
Brief Title: Efficacy and Safety of Bevacizumab Versus Pulvis Talci in Malignant Pleural Effusion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Xiaofei Li, chief physician, Tang-Du Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTSL002
Record Dates: First submitted 2014-01-28; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab (Experimental): Bevacizumab200mg by intrapleural administration
  Interventions: Drug: Bevacizumab
- Pulvis talci (Active Comparator): Pulvis talci 4g by intrapleural administration
  Interventions: Drug: Pulvis talci

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab200mg by intrapleural administration
  Other Names: Avastin
  Arms: Bevacizumab
Drug: Pulvis talci — Pulvis talci 4g by intrapleural administration
  Arms: Pulvis talci

SUMMARY:
Patients with Malignant pleural effusion can be diagnosis advanced cancer. Currently recognized as the most reliable method to control malignant pleural effusion is pleural fixed or thoracic catheter drainage. The most effective pleural fixed agent is pulvis talci, but there are about 30% relapse rate. Thoracic drainage can lead to some complications, such as chest infections, catheter migration and blockage etc. The investigators need a reliable methods to solve dyspnea and other symptoms caused by malignant pleural effusion, and improve quality of life. The purpose of this study was to determine the efficacy and Safety of intrapleural Bevacizumab versus pulvis talci as treatment for malignant pleural effusions (MPE) in patients.

DETAILED DESCRIPTION:
Background： Patients with Malignant pleural effusion can be diagnosis advanced cancer. Currently recognized as the most reliable method to control malignant pleural effusion is pleural fixed or thoracic catheter drainage. The most effective pleural fixed agent is pulvis talci, but there are about 30% relapse rate. Thoracic drainage can lead to some complications, such as chest infections, catheter migration and blockage etc. The investigators need a reliable methods to solve dyspnea and other symptoms caused by malignant pleural effusion, and improve quality of life. The purpose of this study was to determine the efficacy and Safety of intrapleural Bevacizumab versus pulvis talci as treatment for malignant pleural effusions (MPE) in patients.

Methods:

A unblended, randomized study to compare the inhibition of two treatment methods in malignant pleural effusion. Consecutive 183 patients were randomly assigned to two groups, A group is Bevacizumab200mg by intrapleural administration; B group is injected pulvis talci with closed thoracic drainage.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnose malignant pleural effusions by:

   * Diagnose malignant pleural neoplasms by histopathology
   * Recurrent pleural effusion, Histologically or cytologically confirmed diagnosis of cancer
2. Written informed consent

Exclusion Criteria:

1. <18years of age
2. Expected survival <3 months
3. Chest infection, chylothorax, pleurodesis or ipsilateral lung surgery once
4. Planned chemotherapy
5. Pregnancy or breast-feeding (women of child-bearing potential)
6. Not signed informed consent or non-compliance with treatment protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Changes in chest drainage | up to 3months
  Observed chest drainage every day

SECONDARY OUTCOMES:
the average daily VAS defining breathlessness | up to 1 year
  VAS: Visual Analogue Scale
Average daily thoracalgia assessed using VAS score | up to 1 year
  VAS: Visual Analogue Scale
percentage of adverse reactions | up to 1 year
Length of Stay | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China